CLINICAL TRIAL: NCT01202994
Title: Practice Effects and Amyloid Imaging Using 18F-PIB (18F-39-F-6-OH-BTA1) Known as [18FGE067]) or Flutemetamol PET and FDG-PET
Brief Title: Practice Effects and Amyloid Imaging Using 18F-PIB or Flutemetamol PET and FDG-PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 43306
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Results first posted 2018-01-11 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Mild cognitive impairment; PET; Practice effects
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flute (Experimental): Flutemetamol PET scan.
  Interventions: Drug: 18F-Flutemetamol

INTERVENTIONS:
Drug: 18F-Flutemetamol — All subjects will undergo a PET scan with 18F-PIB, within six months of also undergoing an FDG-PET scan (PET scans will occur on separate days).
  For the 18F-PIB PET scan: Approximately 185 MBq (5 mCi) of 18F-PIB will be injected intravenously and PET data collected for each subject.
  The FDG-PET scan will follow the same procedures as routine scans obtained in a clinical setting (approximately 370 MBq of 18F-FDG will be injected intravenously and PET data collected for each subject). FDG-PET data will be used to correlate metabolic changes and for anatomic co-registration of 18F-PIB images.
  Other Names: 18F-39-F-6-OH-BTA1; [18FGE067]; Flutametamol PET

SUMMARY:
Alzheimer's disease (AD) is the most common cause of progressive cognitive decline in the United States. AD is characterized by severe impairments in learning, memory and other cognitive abilities that significantly interfere with daily functioning. The neuropathologic hallmarks of AD consist of neuritic plaques, neurofibrillary tangles, and selective neuronal cell loss. Amyloid plaques, which contain Abeta protein, are believed to play an integral role in the development of AD. Elevated levels of Abeta in the brain are also correlated with cognitive decline.

Alzheimer's (AD) develops insidiously, making it difficult to identify early, yet treatment is most effective when begun during the early stages of the disease. Thus, it has become important for researchers to identify markers of early AD. This project will examine the relationship between four potential markers that may indicate the early development of AD:

1. Mild cognitive impairment (MCI)or normal cognition
2. Practice effects
3. Amyloid plaque binding on 18F-PIB PET
4. Glucose hypometabolism on FDG PET

This project will recruit 25 subjects from an ongoing community-based study of memory and practice effects in cognitively normal, community-dwelling individuals who are age 65 and over (NIA #5K23AG028417-05). Each subject will undergo positron emission tomography (PET) with both 18F-Flutemetamol and FDG.

The overall objective of this companion project is to study the biodistribution and binding of 18F-Flutemetamol in these subjects using PET imaging, which will provide biological evidence to support the overall hypothesis that failure to benefit from practice on a learning paradigm is an early marker of AD.

DETAILED DESCRIPTION:
The overall objective of this companion study project is to study the biodistribution and binding of 18F-Flutemetamol using PET imaging in community-dwelling functionally intact elderly subjects. Understanding the biodistribution and binding of this radiopharmaceutical in normal patients with various levels of potential for cognitive decline will help determine its appropriate role as a disease biomarker and aid in the interpretation of images produced with this agent. Comparison with FDG-PET is essential to correlate metabolic changes and for anatomic co-registration of 18F-PIB images necessary for group analysis.

We will use 18F-Flutemetamol and FDG-PET to compare subjects with low and high practice effects with the following aims and hypotheses:

Specific Aim 1: Examine the relationship between practice effects and amyloid burden in a community sample.

Specific Aim 2: Determine whether FDG-PET or 18F-Flutemetamol better distinguish individuals with high and low practice effects.

Hypothesis 1: Practice effects will be negatively correlated with amyloid deposition, so that higher levels of practice effects (i.e., better repeat testing) will be associated with lower levels of brain amyloid deposition and lower levels of practice effects (i.e., poorer repeat testing) will be associated with greater levels of brain amyloid and these two groups are more clearly distinguishable with 18F-PIB than FDG-PET.

Hypothesis 2: Patients with increased amyloid deposition shown with 18F-PIB will have an FDG-PET scan with more pronounced temporal and parietal hypometabolism as noted on visual review of images and on statistical image analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be currently enrolled in an NIA-sponsored, community-based study of practice effects in non-demented adults age 65 and older living independently (NIA #5K23AG028417-05)

Exclusion Criteria:

* History of neurological disease known to affect cognition (e.g., stroke, head injury with loss of consciousness of >30 minutes, seizure disorder, demyelinating disorder, mental retardation, etc.)
* Dementia based on DSM-IV criteria
* Current or past major psychiatric illness (e.g., schizophrenia, bipolar affective disorder)
* 30-item Geriatric Depression Score >14
* Evidence of stroke or mass lesion on CT or MRI scan
* History of alcoholism or other substance abuse
* Current use of cholinesterase inhibitors, other cognitive enhancers, antipsychotics, or anticonvulsant medications
* History of radiation therapy to the brain
* History of significant major medical illnesses, such as cancer or AIDS
* Uncontrolled diabetes or blood glucose >180 mg/dl on the day of the FDG-PET scan
* Currently pregnant

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Duff, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Center for Alzheimer's Care, Imaging and Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Flute and pe: Participants receive a flutemetamol PET scan and two cognitive testing sessions across one week
Period: Overall Study
Arm/Group | Flute and pe
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Flute and pe
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Amyloid Deposition Obtained on a 18F-flutemetamol Brain Scan.
Description: Standardized Uptake Value Ratio on flutemetamol scan will be the imaging marker of Alzheimer's disease pathology.
Time Frame: Imaging occurred during a single session with each subject.
Measure: Mean (Standard Deviation); unit: ratio of flutemetamol absorbed
Groups:
- Flute: Flutemetamol PET scan.
  18F-Flutemetamol: All subjects will undergo a PET scan with 18F-PIB. Approximately 185 MBq (5 mCi) of 18F-PIB will be injected intravenously and PET data collected for each subject.
Arm/Group | Flute
Number analyzed (Participants) | 27
ratio of flutemetamol absorbed | 1.65 (1.30)
Statistical Analysis 1: Comparison: Flute; The primary analysis is to examine the correlation between the practice effect z-score (presented in the Secondary Outcome section) and the standardized uptake value of flutemetamol (presented in the Outcome module); Test type: Other; p < 0.05, correlation — This is a calculated p-value; correlation coefficient = -0.45

2. Secondary Outcome: Change in Participant Z-score
Description: This z-scores is based on a test of visual learning and memory, which was administered to subjects twice across one week. The amount of change that individuals show across one week is the baseline measure assessed with this variable. We focused on the amount of change observed on the Delayed Recall trial of this test between baseline and one week (i.e., practice effect). The practice effect score on this test is represented as a z-score (M = 0, SD = 1), with higher scores indicating more improvement across one week, which is better result than lower scores.
Time Frame: baseline, one week
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Flute: Flutemetamol PET scan.
  18F-Flutemetamol: All subjects will undergo a PET scan with 18F-PIB, within six months of also undergoing an FDG-PET scan (PET scans will occur on separate days).
  For the 18F-PIB PET scan: Approximately 185 MBq (5 mCi) of 18F-PIB will be injected intravenously and PET data collected for each subject.
  The FDG-PET scan will follow the same procedures as routine scans obtained in a clinical setting (approximately 370 MBq of 18F-FDG will be injected intravenously and PET data collected for each subject). FDG-PET data will be used to correlate metabolic changes and for anatomic co-registration of 18F-PIB images.
Arm/Group | Flute
Number analyzed (Participants) | 27
z-score | -0.07 (0.77)

ADVERSE EVENTS:
Time Frame: 24 hours after scan.
Arm/Group | Flute and pe
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No